CLINICAL TRIAL: NCT01934452
Title: Prospective Study of Complete Remissions Observed With Sunitinib in Patients With Metastatic Renal Cell Carcinoma mRCC)
Brief Title: Prospective Observational Analysis Of CR With Sunitinib Treatment In mRCC Patients
Acronym: APERCU
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: NRA6180080; A6181209 (Other: Alias Study Number)
Record Dates: First submitted 2013-08-02; First posted 2013-09-04 (Estimated); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-01

CONDITIONS: Complete Remission in Renal Cell Carcinoma
Keywords: complete remission
MeSH Terms: conditions — Pathologic Complete Response | interventions — Sunitinib

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood and serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Complete Remission: Complete remission arm in mRCC patients treated with sunitinib.
  Interventions: Drug: sunitinib
- Non Complete Remission: Non complete remission arm in mRCC patients treated with sunitinib.
  Interventions: Drug: sunitinib

INTERVENTIONS:
Drug: sunitinib — 50 mg 4/2 ,oral, once a day 4 weeks on and 2 weeks off for 6 months
  Other Names: Cases
  Groups: Complete Remission
Drug: sunitinib — 50 mg 4/2 ,oral, once a day 4 weeks on and 2 weeks off for 6 months
  Other Names: Controls
  Groups: Non Complete Remission

SUMMARY:
This prospective study will investigate the characteristics of mRCC patients at time of CR in comparison with mRCC patients non on CR treated with Sunitinib, in order to provide some answers/ refection leads to the following questions :

Can we identify blood specificity at time of CR vs non on CR? Shall we distinguish CR with sunitinib alone from combined CR (sunitinib with local treatment), while in clinical report these 2 cohorts present similar time to recurrence (ALBIGES, ASCO 2010)? Can we identify potential predictive serum biomarkers of recurrence? (With the aim of isolating blood biomarker that can help on treatment discontinuation decision?)

DETAILED DESCRIPTION:
The main objective of the study is to describe the characteristics of mRCC patients on CR with Sunitinib (Cases) and compare them to the characteristics of mRCC patients non on CR (controls) in order to identify factors associated with the occurrence of complete remission.

The results obtained on the sample must be representative of the population targeted by the study. The most appropriate method to obtain a representative sample is probability sampling.

A sample size of N = 40 (cases) and N = 80 (Controls) will provide a power of 80% in the detection of a frequency difference between cases and controls corresponding to an OR of 0.24 for a parameter frequency 10% in control arm and an OR of 0.30 for a parameter frequency of around 30% in control arm. The significance level was set at bilateral 5%.

The data will be analyzed using SAS software (version 9.1 - SAS Institute, North Carolina, United States).

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic renal cell carcinoma, histopathologically confirmed
* Treated with sunitinib according to Smpc
* For cases: Achieving a CR (local assessment according to RECIST V1.0 criteria) with Sunitinib in prior 6 months alone OR in combination with local treatment (surgery, radiation therapy, ablative techniques: cryotherapy, RFA)
* For controls: Life expectancy > 3 months No prior Sunitinib treatment
* Patient >18 years

Exclusion Criteria:

* Sunitinib administered in a non-approved label
* For cases: CR occurring without sunitinib treatment
* For controls: Prior systemic treatment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: complete remission in mRCC patients treated with sunitinib versus non complete remission in mRCC patients treated with sunitinib
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2015-05-21 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- France (14):
  - CHU de la Timone, Marseille, Cedex 5
  - CHU Strasbourg, Strasbourg, Cedex
  - CHRU HOTEL DIEU - Service Urologie, Angers
  - C.H.U Morvan, Brest
  - Clinique Victor Hugo, Le Mans
  - Institut Paoli-Calmettes / Hôpital de jour, Marseille
  - Institut Paoli-Calmettes, Marseille
  - Hopital Timone Adultes, Marseille
  - CRLC Val d'Aurelle, Montpellier
  - Hopital Europeen Georges Pompidou, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Clinique Chirurgicale de l'Orangerie, Chiliotherapie, Strasbourg
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=NRA6180080&StudyName=Prospective%20Observational%20Analysis%20Of%20CR%20With%20Sunitinib%20Treatment%20In%20mRCC%20Patients%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants diagnosed with metastatic renal cell carcinoma (mRCC), aged above 18 years treated with sunitinib, were included in this study and their data was observed prospectively.
Groups:
- Sunitinib: Complete Remission (Cases): Participants with mRCC in complete remission treated with sunitinib in real world clinical practice as per summary of product characteristics were included in this reporting arm.
- Sunitinib: Non-Complete Remission (Control): Participants with mRCC in non-complete remission treated with sunitinib in real world clinical practice as per summary of product characteristics were included in this reporting arm.
Period: Overall Study
Arm/Group | Sunitinib: Complete Remission (Cases) | Sunitinib: Non-Complete Remission (Control)
Started | 35 | 42
Completed | 35 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose data were observed in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sunitinib: Complete Remission (Cases) | Sunitinib: Non-Complete Remission (Control) | Total
Number analyzed (Participants) | 35 | 42 | 77
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.5 (9.1) | 60.3 (10.1) | 60.4 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 26 | 31 | 57
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Time to Diagnose Metastatic Renal Cell Carcinoma
Description: Time to diagnose metastatic renal cell carcinoma was defined as the duration between date of diagnosis of mRCC to date of inclusion visit.
Time Frame: Baseline (at inclusion Visit)
Population: Analysis population included all eligible participants whose data were observed in the study.
Measure: Median (Inter-Quartile Range); unit: Years
Arm/Group | Sunitinib: Complete Remission (Cases) | Sunitinib: Non-Complete Remission (Control)
Number analyzed (Participants) | 35 | 42
Years | 3.79 [2.39 to 5.42] | 0.21 [0.09 to 0.82]
Statistical Analysis 1: Comparison: Sunitinib: Complete Remission (Cases) vs Sunitinib: Non-Complete Remission (Control); Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Hodges Lehmann estimator = 2.8, 95% CI 2-sided [2.2 to 3.8]

2. Primary Outcome: Number of Participants Categorized According to Presence of Nephrectomy
Description: In this outcome measure, participants were categorized according to presence of nephrectomy as yes or no.
Time Frame: Baseline (at inclusion Visit)
Population: Analysis population included all eligible participants whose data were observed in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases) | Sunitinib: Non-Complete Remission (Control)
Number analyzed (Participants) | 35 | 42
Participants
  Yes | 35 | 31
  No | 0 | 11
Statistical Analysis 1: Comparison: Sunitinib: Complete Remission (Cases) vs Sunitinib: Non-Complete Remission (Control); Test type: Superiority; p = 0.001, Chi-squared

3. Primary Outcome: Number of Participants Categorized According to Type of Nephrectomy
Description: In this outcome measure, participants were categorized according to type of nephrectomy. Various types of nephrectomies included: extended or partial, nephrectomy with or without adrenalectomy, nephrectomy with or without curettage and open or laparoscopic nephrectomy.
Time Frame: Baseline (at inclusion Visit)
Population: Analysis population included all eligible participants whose data were observed in the study. Here, "Overall number of participants analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable with non-missing values for specific rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases) | Sunitinib: Non-Complete Remission (Control)
Number analyzed (Participants) | 35 | 31
Participants
  Extended or partial nephrectomy: Extended: number analyzed (Participants) | 34 | 31
  Extended or partial nephrectomy: Extended | 30 | 28
  Extended or partial nephrectomy: Partial: number analyzed (Participants) | 34 | 31
  Extended or partial nephrectomy: Partial | 4 | 3
  Nephrectomy with or without adrenalectomy: With adrenalectomy: number analyzed (Participants) | 33 | 26
  Nephrectomy with or without adrenalectomy: With adrenalectomy | 15 | 11
  Nephrectomy with or without adrenalectomy: Without adrenalectomy: number analyzed (Participants) | 33 | 26
  Nephrectomy with or without adrenalectomy: Without adrenalectomy | 18 | 15
  Nephrectomy with or without curettage: With curettage: number analyzed (Participants) | 32 | 25
  Nephrectomy with or without curettage: With curettage | 11 | 2
  Nephrectomy with or without curettage: Without curettage: number analyzed (Participants) | 32 | 25
  Nephrectomy with or without curettage: Without curettage | 21 | 23
  Open or laparoscopic nephrectomy: Laparoscopic nephrectomy: number analyzed (Participants) | 26 | 21
  Open or laparoscopic nephrectomy: Laparoscopic nephrectomy | 5 | 5
  Open or laparoscopic nephrectomy: Open nephrectomy: number analyzed (Participants) | 26 | 21
  Open or laparoscopic nephrectomy: Open nephrectomy | 21 | 16
Statistical Analysis 1: Comparison: Sunitinib: Complete Remission (Cases) vs Sunitinib: Non-Complete Remission (Control); Extended or partial nephrectomy; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 2: Comparison: Sunitinib: Complete Remission (Cases) vs Sunitinib: Non-Complete Remission (Control); Nephrectomy with or without adrenalectomy; Test type: Superiority; p = 0.809, Chi-squared
Statistical Analysis 3: Comparison: Sunitinib: Complete Remission (Cases) vs Sunitinib: Non-Complete Remission (Control); Nephrectomy with or without curettage; Test type: Superiority; p = 0.019, Chi-squared
Statistical Analysis 4: Comparison: Sunitinib: Complete Remission (Cases) vs Sunitinib: Non-Complete Remission (Control); Open or laparoscopic nephrectomy; Test type: Superiority; p = 0.734, Fisher Exact

4. Primary Outcome: Time to Nephrectomy From Diagnosis of Metastatic Renal Cell Carcinoma (mRCC)
Description: In this outcome measure, time from diagnosis of mRCC to nephrectomy was reported.
Time Frame: Baseline (at inclusion Visit)
Population: Analysis population included all eligible participants whose data were observed in the study. Here, "Overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Sunitinib: Complete Remission (Cases) | Sunitinib: Non-Complete Remission (Control)
Number analyzed (Participants) | 33 | 28
Months | 5.7 [-0.5 to 20.3] | 10.0 [-0.4 to 29.6]
Statistical Analysis 1: Comparison: Sunitinib: Complete Remission (Cases) vs Sunitinib: Non-Complete Remission (Control); Test type: Superiority; p = 0.230, Wilcoxon (Mann-Whitney); Hodges Lehmann estimator = -3.7, 95% CI 2-sided [-13.2 to 1.6]

5. Primary Outcome: Number of Participants Categorized According to Pathological Classification
Description: In this outcome measure, participants were categorized according to pathological classification. Pathological classification included: clear cell carcinoma (yes or no), multilocular cystic renal clear cell carcinoma (yes or no), papillary cell carcinoma (yes or no), chromophobe cell carcinoma(yes or no), Bellini's collecting duct carcinoma(yes or no), medullary cell carcinoma (yes or no), sarcomatoid contingent (yes or no), and other (yes or no).
Time Frame: Baseline (at inclusion Visit)
Population: Analysis population included all eligible participants whose data were observed in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases) | Sunitinib: Non-Complete Remission (Control)
Number analyzed (Participants) | 35 | 42
Participants
  Clear cell carcinoma: Yes | 33 | 39
  Clear cell carcinoma: No | 2 | 3
  Multilocular cystic renal clear cell carcinoma: Yes | 1 | 1
  Multilocular cystic renal clear cell carcinoma: No | 34 | 41
  Papillary cell carcinoma: Yes | 1 | 4
  Papillary cell carcinoma: No | 34 | 38
  Chromophobe cell carcinoma: Yes | 1 | 0
  Chromophobe cell carcinoma: No | 34 | 42
  Bellini's collecting duct carcinoma: Yes | 0 | 1
  Bellini's collecting duct carcinoma: No | 35 | 41
  Medullary cell carcinoma: Yes | 0 | 0
  Medullary cell carcinoma: No | 35 | 42
  Sarcomatoid contingent: Yes | 4 | 3
  Sarcomatoid contingent: No | 31 | 39
  Other: Yes | 3 | 2
  Other: No | 32 | 40
Statistical Analysis 1: Comparison: Sunitinib: Complete Remission (Cases) vs Sunitinib: Non-Complete Remission (Control); Sarcomatoid contingent; Test type: Superiority; p = 0.695, Fisher Exact

6. Primary Outcome: Number of Participants Categorized According to Tumor, Node, Metastasis (TNM) Classification
Description: In this outcome measure, participants were categorized according to TNM classification. TNM classification included: T class (1, 2, 3, 4), N (0,1,2, x) and M class (0, 1). TNM system is based on size of primary tumor (T), amount of spread to lymph nodes (N) and presence of metastases (M). T1: tumor (less than or equal to) <=20 millimeters (mm), T2: tumor >20 mm to <=50 mm, T3: >50 mm, T4: tumor invading other structures. N0: no lymph node metastases, N1: metastases to ipsilateral level I, II axillary lymph nodes, NX: Regional lymph nodes cannot be assessed. M0: no clinical/radiographic evidence of distant metastases, M1: distant detectable metastases as determined by clinical and radiographic means and/or histologically proven >0.2 mm.
Time Frame: Baseline (at inclusion Visit)
Population: Analysis population included all eligible participants whose data were observed in the study. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable with non-missing value for specific rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases) | Sunitinib: Non-Complete Remission (Control)
Number analyzed (Participants) | 34 | 34
Participants
  T Class: T1 | 8 | 8
  T Class: T2 | 7 | 8
  T Class: T3 | 18 | 15
  T Class: T4 | 1 | 3
  N Class: N0: number analyzed (Participants) | 23 | 21
  N Class: N0 | 12 | 10
  N Class: N1: number analyzed (Participants) | 23 | 21
  N Class: N1 | 1 | 3
  N Class: N2: number analyzed (Participants) | 23 | 21
  N Class: N2 | 2 | 2
  N Class: NX: number analyzed (Participants) | 23 | 21
  N Class: NX | 8 | 6
  M Class: M0: number analyzed (Participants) | 32 | 32
  M Class: M0 | 19 | 15
  M Class: M1: number analyzed (Participants) | 32 | 32
  M Class: M1 | 13 | 17
Statistical Analysis 1: Comparison: Sunitinib: Complete Remission (Cases) vs Sunitinib: Non-Complete Remission (Control); M class; Test type: Superiority; p = 0.316, Chi-squared

7. Primary Outcome: Tumour Size
Description: Tumour size of participants was reported in this outcome measure.
Time Frame: Baseline (at Inclusion Visit)
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: Millimeter
Arm/Group | Sunitinib: Complete Remission (Cases) | Sunitinib: Non-Complete Remission (Control)
Number analyzed (Participants) | 34 | 34
Millimeter | 73.0 [48.0 to 110.0] | 75.5 [50.0 to 100.0]
Statistical Analysis 1: Comparison: Sunitinib: Complete Remission (Cases) vs Sunitinib: Non-Complete Remission (Control); Test type: Superiority; p = 0.778, Wilcoxon (Mann-Whitney); Hodges Lehmann estimator = -2.0, 95% CI 2-sided [-22.0 to 18.0]

8. Primary Outcome: Number of Participants Categorized According to Fuhrman Nuclear Grade
Description: In this outcome measure, participants were categorized according to Fuhrman nuclear grade. The grades were classified as: grade 1, 2, 3, and 4. The four-tiered Fuhrman grading evaluates nuclear size, nuclear shape and presence of nucleolar prominence. Grade 1: small (=10 micrometer [mcm]) nuclear diameter, round/uniform nuclear shape and absent/inconspicuous nucleoli; Grade 2: large (=15 mcm) nuclear diameter, irregular outline nuclear shape and visible at *400 magnification nucleoli; Grade 3: larger (=20 mcm) nuclear diameter, obvious irregular outline nuclear shape and visible and prominent at *100 magnification nucleoli; Grade 4: grade 3 plus bizarre multilobed nuclei +/- spindle cells.
Time Frame: Baseline (at Inclusion Visit)
Population: Analysis population included all eligible participants whose data were observed in the study. Here, "Overall number of participants analyzed" signifies participants evaluable for this outcome measure with non-missing values.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases) | Sunitinib: Non-Complete Remission (Control)
Number analyzed (Participants) | 33 | 34
Participants
  Grade 1 | 2 | 4
  Grade 2 | 9 | 11
  Grade 3 | 14 | 12
  Grade 4 | 8 | 7
Statistical Analysis 1: Comparison: Sunitinib: Complete Remission (Cases) vs Sunitinib: Non-Complete Remission (Control); Test type: Superiority; p = 0.812, Fisher Exact

9. Primary Outcome: Number of Participants Categorized According to Presence of Necrosis, Pulmonary Embolism and Sarcomatoid Component
Description: In this outcome measure, participants were categorized according to presence of necrosis, pulmonary embolism and sarcomatoid component.
Time Frame: Baseline (at Inclusion Visit)
Population: Analysis population included all eligible participants whose data were observed in the study. Here, "Overall number of participants analyzed" signifies participants evaluable for this outcome measure with non-missing values and "number analyzed" signifies participants evaluable at specific rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases) | Sunitinib: Non-Complete Remission (Control)
Number analyzed (Participants) | 34 | 33
Participants
  Presence of necrosis: number analyzed (Participants) | 33 | 31
  Presence of necrosis: Yes | 14 | 20
  Presence of necrosis: No | 19 | 11
  Vascular embolism: number analyzed (Participants) | 32 | 28
  Vascular embolism: Yes | 12 | 12
  Vascular embolism: No | 20 | 16
  Sarcomatoid component: Yes | 5 | 5
  Sarcomatoid component: No | 29 | 28
Statistical Analysis 1: Comparison: Sunitinib: Complete Remission (Cases) vs Sunitinib: Non-Complete Remission (Control); Presence of necrosis; Test type: Superiority; p = 0.077, Chi-squared; Odds Ratio (OR) = 2.47, 95% CI 2-sided [0.90 to 6.77]
Statistical Analysis 2: Comparison: Sunitinib: Complete Remission (Cases) vs Sunitinib: Non-Complete Remission (Control); Vascular embolism; Test type: Superiority; p = 0.673, Chi-squared; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.44 to 3.52]
Statistical Analysis 3: Comparison: Sunitinib: Complete Remission (Cases) vs Sunitinib: Non-Complete Remission (Control); Sarcomatoid component; Test type: Superiority; p = 1.000, Fisher Exact; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.27 to 3.97]

10. Primary Outcome: Time to Initiation of Sunitinib From Diagnosis of Metastatic Renal Cell Carcinoma (mRCC)
Time Frame: Diagnosis of mRCC to Sunitinib Initiation (at Inclusion Visit)
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Sunitinib: Complete Remission (Cases) | Sunitinib: Non-Complete Remission (Control)
Number analyzed (Participants) | 33 | 39
Months | 3.25 [1.54 to 6.47] | 2.69 [1.81 to 9.82]
Statistical Analysis 1: Comparison: Sunitinib: Complete Remission (Cases) vs Sunitinib: Non-Complete Remission (Control); Test type: Superiority; p = 0.865, Wilcoxon (Mann-Whitney); Hodges Lehmann estimator = -0.2, 95% CI 2-sided [-1.5 to 1.6]

11. Primary Outcome: Number of Participants Categorized According to Location of Metastases
Description: In this outcome measure, participants were categorized according to location of metastases at different body parts (lung, bones, liver, adrenal gland, pancreas, brain and lymph nodes). Participant can have more than 1 location of metastases.
Time Frame: At initiation of sunitinib (at Inclusion Visit)
Population: Analysis population included all eligible participants whose data were observed in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases) | Sunitinib: Non-Complete Remission (Control)
Number analyzed (Participants) | 35 | 42
Participants
  Lung: Yes | 15 | 30
  Lung: No | 20 | 12
  Bones: Yes | 5 | 12
  Bones: No | 30 | 30
  Liver: Yes | 6 | 10
  Liver: No | 29 | 32
  Adrenal glands: Yes | 2 | 8
  Adrenal glands: No | 33 | 34
  Pancreas: Yes | 2 | 5
  Pancreas: No | 33 | 37
  Brain: Yes | 0 | 3
  Brain: No | 35 | 39
  Lymph nodes: Yes | 11 | 23
  Lymph nodes: No | 24 | 19
Statistical Analysis 1: Comparison: Sunitinib: Complete Remission (Cases) vs Sunitinib: Non-Complete Remission (Control); Lung; Test type: Superiority; p = 0.011, Chi-squared
Statistical Analysis 2: Comparison: Sunitinib: Complete Remission (Cases) vs Sunitinib: Non-Complete Remission (Control); Bones; Test type: Superiority; p = 0.132, Chi-squared
Statistical Analysis 3: Comparison: Sunitinib: Complete Remission (Cases) vs Sunitinib: Non-Complete Remission (Control); Liver; Test type: Superiority; p = 0.473, Chi-squared
Statistical Analysis 4: Comparison: Sunitinib: Complete Remission (Cases) vs Sunitinib: Non-Complete Remission (Control); Adrenal glands; Test type: Superiority; p = 0.101, Fisher Exact
Statistical Analysis 5: Comparison: Sunitinib: Complete Remission (Cases) vs Sunitinib: Non-Complete Remission (Control); Pancreas; Test type: Superiority; p = 0.445, Fisher Exact
Statistical Analysis 6: Comparison: Sunitinib: Complete Remission (Cases) vs Sunitinib: Non-Complete Remission (Control); Lymph nodes; Test type: Superiority; p = 0.040, Chi-squared

12. Primary Outcome: Number of Participants Categorized According to Type of Lymph Nodes as Metastatic Site
Description: In this outcome measure, participants were categorized according to type of lymph nodes as metastatic site.
Time Frame: At initiation of sunitinib (at Initiation Visit)
Population: Analysis population included all eligible participants whose data were observed in the study. Here, "Overall number of participants analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable at specific rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases) | Sunitinib: Non-Complete Remission (Control)
Number analyzed (Participants) | 11 | 23
Participants
  Supradiaphragmatic: number analyzed (Participants) | 10 | 23
  Supradiaphragmatic: Yes | 7 | 16
  Supradiaphragmatic: No | 3 | 7
  Infradiaphragmatic: Yes | 3 | 11
  Infradiaphragmatic: No | 8 | 12
Statistical Analysis 1: Comparison: Sunitinib: Complete Remission (Cases) vs Sunitinib: Non-Complete Remission (Control); Supradiaphragmatic; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 2: Comparison: Sunitinib: Complete Remission (Cases) vs Sunitinib: Non-Complete Remission (Control); Infradiaphragmatic; Test type: Superiority; p = 0.295, Fisher Exact

13. Primary Outcome: Number of Participants Categorized According to Recurrence at Nephrectomy Site
Description: In this outcome measure, participants were categorized according to recurrence at nephrectomy site were reported.
Time Frame: At initiation of sunitinib (at Inclusion Visit)
Population: Analysis population included all eligible participants whose data were observed in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases) | Sunitinib: Non-Complete Remission (Control)
Number analyzed (Participants) | 35 | 42
Participants
  Yes | 6 | 1
  No | 29 | 41
Statistical Analysis 1: Comparison: Sunitinib: Complete Remission (Cases) vs Sunitinib: Non-Complete Remission (Control); Test type: Superiority; p = 0.042, Fisher Exact

14. Primary Outcome: Number of Participants Categorized According to Recurrence at Other Site
Description: In this outcome measure, participants were categorized according to recurrence at any other site than nephrectomy site were reported.
Time Frame: At initiation of sunitinib (at Inclusion Visit)
Population: Analysis population included all eligible participants whose data were observed in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases) | Sunitinib: Non-Complete Remission (Control)
Number analyzed (Participants) | 35 | 42
Participants
  Yes | 3 | 12
  No | 32 | 30
Statistical Analysis 1: Comparison: Sunitinib: Complete Remission (Cases) vs Sunitinib: Non-Complete Remission (Control); Test type: Superiority; p = 0.027, Chi-squared

15. Primary Outcome: Number of Metastatic Sites
Description: In this outcome measure, median of metastatic sites were reported.
Time Frame: At initiation of sunitinib (at Initiation Visit)
Population: Analysis population included all eligible participants whose data were observed in the study.
Measure: Median (Inter-Quartile Range); unit: Metastatic sites
Arm/Group | Sunitinib: Complete Remission (Cases) | Sunitinib: Non-Complete Remission (Control)
Number analyzed (Participants) | 35 | 42
Metastatic sites | 1.0 [1.0 to 2.0] | 2.0 [2.0 to 4.0]
Statistical Analysis 1: Comparison: Sunitinib: Complete Remission (Cases) vs Sunitinib: Non-Complete Remission (Control); Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Hodges Lehmann estimator = -1.0, 95% CI 2-sided [-1.0 to -1.0]

16. Primary Outcome: Number of Participants Categorized According to Memorial Sloan-Kettering Cancer Center (MSKCC) Prognostic Classification
Description: In this outcome measure, participants were categorized according MSKCC prognostic classification. MSKCC criteria had 5 risk factors: Karnofsky performance status (KPS) <80% (ability to perform ordinary tasks, 0 [dead] -100 [normal]); time from diagnosis to start of systemic therapy <12 months; hemoglobin <lower limit of normal (LLN); lactate dehydrogenase >1.5*upper limit of normal (ULN); corrected serum calcium >10 milligram per deciliter (mg/dL). Present risk factors were added, and participants were stratified as: good prognosis (0 factor), intermediate prognosis (1-2 factors), poor prognosis (>=2 factors).
Time Frame: At initiation of sunitinib (at Inclusion Visit)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases) | Sunitinib: Non-Complete Remission (Control)
Number analyzed (Participants) | 26 | 38
Participants
  Good prognosis | 14 | 8
  Intermediate prognosis | 12 | 24
  Poor prognosis | 0 | 6
Statistical Analysis 1: Comparison: Sunitinib: Complete Remission (Cases) vs Sunitinib: Non-Complete Remission (Control); Test type: Superiority; p = 0.009, Fisher Exact

17. Primary Outcome: Time to Achieve Complete Remission (CR) After Sunitinib Initiation: mRCC Participants With CR
Description: In this outcome measure, time taken by participants to achieve the complete remission after sunitinib initiation were reported. As per Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 criteria: CR = disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to size of <10 millimeter (mm).
Time Frame: From initiation of sunitinib till CR (data collected at Inclusion Visit)
Population: Analysis population included all eligible participants whose data were observed in the study. This outcome measure was planned to be analyzed only in those participants with mRCC in CR.
Measure: Median (Inter-Quartile Range); unit: Years
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 35
Years | 0.98 [-0.8 to 8.0]

18. Primary Outcome: Number of Participants Categorized According to Method of Achieving CR: mRCC Participants With CR
Description: In this outcome measure, participants were categorized according to the method of achieving the CR. Different methods included: treatment combined with local treatment and medical treatment alone. As per RECIST version 1.1 criteria: CR = disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumour marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).
Time Frame: From initiation of sunitinib till CR (data collected at Inclusion Visit)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 35
Participants
  Treatment combined with local treatment | 14
  Medical treatment alone | 21

19. Primary Outcome: Number of Participants Categorized According to Type of Medical Treatment Alone: mRCC Participants With CR
Description: In this outcome measure, participants were categorized according to the type of medical treatment alone as method of achieving the CR. Medical treatment alone included: surgery, radiotherapy, radiofrequency, cryoablation and metastasectomy. Only those categories in which at least 1 participant had data were reported. Participant could have received more than 1 type of medical treatment. As per RECIST version 1.1 criteria: CR = disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumour marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).
Time Frame: From initiation of sunitinib till CR (data collected at Inclusion Visit)
Population: Analysis population included all eligible participants whose data were observed in the study. Here, "Overall number of participants analyzed" signifies participants evaluable for this outcome measure. This outcome measure was planned to be analyzed only in those participants with mRCC in CR.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 14
Participants
  Surgery | 5
  Radiotherapy | 2
  Radiofrequency | 2
  Metastasectomy | 8
  Other | 3

20. Primary Outcome: Number of Participants Categorized According to Treatment Combined With Local Treatment: mRCC Participants With CR
Description: In this outcome measure, participants were categorized according to the type of treatment Combined With local treatment alone as method of achieving the CR. Type of treatment combined with local treatment included: surgery, surgery + radiotherapy + radiofrequency + metastasectomy, metastasectomy, metastasectomy + other, radiofrequency + metastasectomy + other and radiotherapy. As per RECIST version 1.1 criteria: CR = disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumour marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).
Time Frame: From initiation of sunitinib till CR (data collected at Inclusion Visit)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 14
Participants
  Other | 1
  Surgery | 4
  Surgery + Radiotherapy + Radiofrequency + Metastasectomy | 1
  Metastasectomy | 5
  Metastasectomy + Other | 1
  Radiofrequency + Metastasectomy + Other | 1
  Radiotherapy | 1

21. Primary Outcome: Number of Participants Categorized According to Radiological Assessment of the CR: mRCC Participants With CR
Description: In this outcome measure, participants were categorized according to radiological assessment of the CR. It included: disappearance of all known target lesions, disappearance of all non-target lesions, no new lesions and all target and non-target lymph nodes. Only those categories with at least 1 participant as result are reported. As per RECIST version 1.1 criteria: CR = disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumour marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).
Time Frame: From initiation of sunitinib till CR (data collected at Inclusion Visit)
Population: Analysis population included all eligible participants whose data were observed in the study. Here, "number analyzed" signifies participants evaluable with non-missing values for specified rows. This outcome measure was planned to be analyzed only in those participants with mRCC in CR.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 35
Participants
  Disappearance of all known target lesions: yes | 35
  Disappearance of all non-target lesions: yes: number analyzed (Participants) | 34
  Disappearance of all non-target lesions: yes | 34
  No new lesions: yes | 34
  No new lesions: no | 1
  All target and non-target lymph nodes: yes: number analyzed (Participants) | 34
  All target and non-target lymph nodes: yes | 34

22. Primary Outcome: Number of Participants Categorized According to Therapeutic Strategy After CR: mRCC Participants With CR
Description: In this outcome measure, participants were categorized according to therapeutic strategy after CR. As per RECIST version 1.1 criteria: CR = disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumour marker level. All lymph nodes must be non-pathological in size (<10 mm short axis). It included discontinuation and continuation of sunitinib treatment.
Time Frame: After achieving CR with sunitinib treatment (data collected at Inclusion Visit)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 35
Participants
  Discontinuation of Sunitinib treatment | 16
  Continuation of Sunitinib treatment | 19

23. Primary Outcome: Number of Participants With Disease Evolution (DE) at Month 12 Follow-up Visit: mRCC Participants With CR
Description: DE included:complete response, progression, stabilization and not assessed. Disease progression (PD):per RECIST v1.1: at least 20% increase in sum of diameters of target lesions,taking as reference smallest sum on study.In addition to relative increase of 20%, sum must also demonstrate an absolute increase of at least 5mm.Appearance of 1 or more new lesions was also considered progression. CR:disappearance of all target lesions.Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis) and stable disease (SD): absence of sufficient reduction for a partial response (PR): at least 30% decrease in sum of diameters of target lesions, taking as reference baseline sum diameters or absence of a sufficient increase for PD, taking as reference the sum of lowest diameters during study.
Time Frame: Month 12 follow-up visit
Population: Analysis population included all eligible participants whose data were observed in the study and who had attended at least Month 12 follow-up visit. Here, "Overall number of participants analyzed" signifies participants evaluable for this outcome measure with non-missing values. This outcome measure was planned to be analyzed only in those participants with mRCC in CR.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 31
Participants
  Complete response | 21
  Progression | 5
  Stabilization | 3
  Not assessed | 2

24. Primary Outcome: Number of Participants With Ongoing Sunitinib Treatment at Month 12 Follow-up Visit: mRCC Participants With CR
Description: In this outcome measure, participants with ongoing sunitinib treatment were reported.
Time Frame: Month 12 follow-up study visit
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 29
Participants
  Yes | 9
  No | 20

25. Primary Outcome: Number of Participants With Ongoing Sunitinib Treatment According to Dose and Regimen at Month 12 Follow-up Visit: mRCC Participants With CR
Description: In this outcome measure, participants with ongoing sunitinib treatment according to dose (25, 37.5 and 50 mg) and regimen (4/2 [4 weeks dosing then 2 weeks off] and 2/1 [4 weeks dosing then 2 weeks off]) were reported.
Time Frame: Month 12 follow-up study visit
Population: Analysis population included all eligible participants whose data were observed in the study and who had attended at least Month 12 follow-up visit. Here, "Overall number of participants analyzed" signifies participants evaluable for this outcome measure. This outcome measure was planned to be analyzed only in those participants with mRCC in CR.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 9
Participants
  Current dose: 25 mg | 1
  Current dose: 37.5 mg | 4
  Current dose: 50 mg | 4
  Current regimen: 4/2 | 1
  Current regimen: 2/1 | 6
  Current regimen: other | 2

26. Primary Outcome: Number of Participants Who Discontinued Sunitinib Temporarily at Month 12 Follow-up Visit: mRCC Participants With CR
Description: In this outcome measure, participants who temporarily discontinued sunitinib were reported.
Time Frame: Month 12 follow-up study visit
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 26
Participants
  Yes | 5
  No | 21

27. Primary Outcome: Number of Participants Categorized According to Number of Temporary Discontinuations of Sunitinib Treatment at Month 12 Follow-up Visit: mRCC Participants With CR
Description: In this outcome measure, participants were categorized according to number (1 and 2) of temporary discontinuations of sunitinib.
Time Frame: Month 12 follow-up study visit
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 5
Participants
  1-time temporary discontinuation | 3
  2-times temporary discontinuation | 2

28. Primary Outcome: Number of Instances When Different Types of Reason Led to Temporary Discontinuation of Sunitinib Treatment at Month 12 Follow up Visit: mRCC Participants With CR
Description: In this outcome measure, number of instances when different types of reasons led to temporary discontinuations like intolerance, local treatment and other reasons were reported. Participant could have temporarily discontinued sunitinib treatment more than once.
Time Frame: Month 12 follow-up study visit
Population: as for outcome 25
Measure: Number; unit: Instances
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 5
Instances
  Intolerance | 3
  Local treatment | 1
  Others | 3

29. Primary Outcome: Number of Instances When Participants Resumed Sunitinib Treatment After Temporary Discontinuation at Month 12: mRCC Participants With CR
Description: In this outcome measure, number of instances when participants resumed sunitinib treatment were reported. Participant could have temporarily discontinued sunitinib treatment more than once and likewise resumed treatment more than once.
Time Frame: Month 12 follow-up study visit
Population: as for outcome 25
Measure: Number; unit: Instances
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 5
Instances
  Resumed: yes | 6
  Resumed: no | 1

30. Primary Outcome: Duration of Temporary Discontinuation of Sunitinib Treatment at Month 12 Follow-up Visit: mRCC Participants With CR
Description: In this outcome measure, duration of temporary discontinuation of sunitinib treatment were reported.
Time Frame: Month 12 follow-up study visit
Population: as for outcome 25
Measure: Median (Full Range); unit: Days
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 5
Days | 15.0 [4 to 93]

31. Primary Outcome: Number of Participants Who Discontinued Sunitinib Permanently at Month 12 Follow-up Visit: mRCC Participants With CR
Description: In this outcome measure, number of participants who permanently discontinued sunitinib were reported.
Time Frame: Month 12 follow-up study visit
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 27
Participants
  Yes | 10
  No | 17

32. Primary Outcome: Number of Participants Categorized According to Reasons for Permanent Discontinuations of Sunitinib Treatment at Month 12 Follow-up Visit: mRCC Participants With CR
Description: In this outcome measure, participants were categorized according to reasons for permanent discontinuation of sunitinib.
Time Frame: Month 12 follow-up visit
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 10
Participants
  Intolerance | 1
  Complete response retention | 7
  Decision of participant or doctor | 1
  Other | 1

33. Primary Outcome: Duration of Treatment With Sunitinib Since Complete Remission at Month 12 Follow-up Visit: mRCC Participants With CR
Description: In this outcome measure, duration of treatment with sunitinib since complete remission was reported.
Time Frame: Month 12 follow-up study visit
Population: as for outcome 25
Measure: Median (Full Range); unit: Months
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 8
Months | 6.00 [0.0 to 37.1]

34. Primary Outcome: Number of Participants With Disease Evolution at Month 24 Follow-up Visit: mRCC Participants With CR
Description: DE included: CR, PD, SD and not assessed. PD: per RECIST v1.1: at least a 20% increase in sum of diameters of target lesions, taking as reference smallest sum on study. In addition to relative increase of 20%, sum must also demonstrate an absolute increase of at least 5mm. Appearance of one or more new lesions was also considered progression. CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).SD: absence of sufficient reduction for PR: at least 30% decrease in sum of diameters of target lesions, taking as reference baseline sum diameters or absence of a sufficient increase for PD, taking as reference the sum of lowest diameters during study.
Time Frame: Month 24 follow-up study visit
Population: Analysis population included all eligible participants whose data were observed in the study and who had attended at least Month 24 follow-up visit. Here, "Overall number of participants analyzed" signifies participants evaluable for this outcome measure with non-missing values. This outcome measure was planned to be analyzed only in those participants with mRCC in CR.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 26
Participants
  Complete response | 19
  Progression | 4
  Stabilization | 1
  Not assessed | 2

35. Primary Outcome: Number of Participants With Ongoing Sunitinib Treatment at Month 24 Follow-up Visit: mRCC Participants With CR
Description: In this outcome measure, participants with ongoing sunitinib treatment were reported.
Time Frame: Month 24 follow-up study visit
Population: Analysis population included all eligible participants whose data were observed in the study and who had attended at least Month 24 follow-up visit. Here, "Overall number of participants analyzed" signifies participants evaluable for this outcome measure. This outcome measure was planned to be analyzed only in those participants with mRCC in CR.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 25
Participants
  Yes | 4
  No | 21

36. Primary Outcome: Number of Participants Who Discontinued Sunitinib Temporarily at Month 24 Follow-up Visit: mRCC Participants With CR
Description: In this outcome measure, number of participants who temporarily discontinued sunitinib were reported.
Time Frame: Month 24 follow-up study visit
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 23
Participants
  Yes | 2
  No | 21

37. Primary Outcome: Number of Participants Who Resumed Treatment at Month 24 Follow-up Visit: mRCC Participants With CR
Description: In this outcome measure, participants who resumed sunitinib were reported.
Time Frame: Month 24 follow-up study visit
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 1
Participants | 1

38. Primary Outcome: Number of Days of Temporary Discontinuation of Sunitinib Treatment at Month 24 Follow-up Visit: mRCC Participants With CR
Time Frame: Month 24 follow-up study visit
Population: as for outcome 35
Measure: Number; unit: Days
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 1
Days | 15

39. Primary Outcome: Number of Participants Who Discontinued Sunitinib Permanently at Month 24 Follow-up Visit: mRCC Participants With CR
Time Frame: Month 24 follow-up study visit
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 23
Participants
  Yes | 11
  No | 12

40. Primary Outcome: Number of Participants Categorized According to Reasons for Permanent Discontinuations of Sunitinib Treatment at Month 24 Follow-up Visit: mRCC Participants With CR
Time Frame: Month 24 follow-up study visit
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 11
Participants
  Progression | 1
  Intolerance | 3
  Complete response retention | 7

41. Primary Outcome: Duration of Treatment With Sunitinib Since Complete Remission at Month 24 Follow-up Visit: mRCC Participants With CR
Description: CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).
Time Frame: Month 24 follow-up study visit
Population: as for outcome 35
Measure: Median (Full Range); unit: Months
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 9
Months | 7.62 [0.0 to 37.1]

42. Primary Outcome: Time to Progression With Sunitinib Treatment From Complete Remission: mRCC Participants With CR
Description: CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis). PD: =>20% increase in sum of longest dimensions of lesions taking as a reference smallest sum of longest dimensions since treatment start or appearance of =>1 new lesions.
Time Frame: From achieving CR with Sunitinib treatment (before inclusion in the study, participants recruited for 3 years) to Visit at progression (during study); [post inclusion follow-up in the study was maximum of 39.8 months for Cases]
Population: as for outcome 35
Measure: Median (Full Range); unit: Months
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 19
Months | 12.65 [2.0 to 51.8]

43. Primary Outcome: Duration of Additional Treatment With Sunitinib Since Complete Remission: mRCC Participants With CR
Description: as for outcome 41
Time Frame: From complete remission (before inclusion in the study, participants recruited for 3 years) till discontinuation of additional treatment during this study; [post inclusion follow-up in the study was maximum of 39.8 months for Cases]
Population: as for outcome 19
Measure: Median (Full Range); unit: Months
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 11
Months | 10.0 [2 to 49]

44. Primary Outcome: Number of Participants Categorized According to Types of Progression: mRCC Participants With CR
Description: As per RECIST version 1.1, PD was defined as at least a 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered progression.
Time Frame: Study visit at progression; post inclusion follow-up in the study was maximum of 39.8 months for Cases
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 19
Participants
  Local progression | 1
  Distant progression | 18

45. Primary Outcome: Number of Participants Categorized According to Site of Progression: mRCC Participants With CR
Description: as for outcome 44
Time Frame: Study visit at progression; post inclusion follow-up in the study was maximum of 39.8 months for Cases
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 19
Participants
  Known metastatic site: Yes | 12
  Known metastatic site: No | 7
  New metastatic site: Yes | 12
  New metastatic site: No | 7

46. Primary Outcome: Number of Participants Categorized According to Location of Metastases: mRCC Participants With CR
Description: In this outcome measure, participants were categorized according to location of metastases at different body parts (lung, bones, liver, adrenal glands, pancreas, brain, lymph nodes, recurrence at nephrectomy site and other). Participant could have more than 1 location of metastases.
Time Frame: Study visit at progression; post inclusion follow-up in the study was maximum of 39.8 months for Cases
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 19
Participants
  Lung | 7
  Bones | 4
  Liver | 0
  Adrenal glands | 1
  Pancreas | 2
  Brain | 2
  Lymph nodes | 5
  Recurrence at nephrectomy site | 1
  Other | 2

47. Primary Outcome: Number of Participants Categorized According to Type of Lymph Nodes as Metastatic Site: mRCC Participants With CR
Description: In this outcome measure, participants were categorized according to type of lymph nodes as metastatic site were reported.
Time Frame: Study visit at progression; post inclusion follow-up in the study was maximum of 39.8 months for Cases
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 5
Participants
  Supradiaphragmatic: Yes | 3
  Supradiaphragmatic: No | 2
  Infradiaphragmatic: Yes | 2
  Infradiaphragmatic: No | 3

48. Primary Outcome: Number of Participants Categorized According to Number of Metastatic Sites: mRCC Participants With CR
Description: In this outcome measure, participants were categorized according to number of metastatic sites (1, 2 and 3).
Time Frame: Study visit at progression; post inclusion follow-up in the study was maximum of 39.8 months for Cases
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 19
Participants
  1 | 14
  2 | 4
  3 | 1

49. Primary Outcome: Number of Participants Who Received Systemic Treatment After Progression: mRCC Participants With CR
Description: In this outcome measure, participants who received systemic treatment after progression were reported.
Time Frame: After progression, during follow up period maximum of 39.8 months for Cases
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 19
Participants
  Yes | 16
  No | 3

50. Primary Outcome: Number of Participants Categorized According to Type of Systemic Treatment Received After Progression: mRCC Participants With CR
Description: In this outcome measure, participants who received systemic treatment after progression were categorized according to type of treatment. Different types of treatment were tyrosine kinase inhibitor- sunitinib restart, radiotherapy and other systemic treatment. Participant could have more than 1 type of treatment.
Time Frame: After progression, during follow up period maximum of 39.8 months for Cases
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 16
Participants
  Tyrosine kinase inhibitor - Sunitinib restart | 11
  Radiotherapy | 6
  Other systemic treatment | 3

51. Primary Outcome: Number of Participants With Best Objective Response After Progression: mRCC Participants With CR
Description: Participants with best objective response after progression were evaluated here. It included complete, partial, stabilized and not applicable. PD per RECIST v1.1: at least a 20% increase in sum of diameters of target lesions,taking as reference smallest sum on study. In addition to relative increase of 20%, sum must also demonstrate an absolute increase of at least 5mm. Appearance of one or more new lesions was also considered progression. CR:disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis) & SD: absence of sufficient reduction for a PR: at least 30% decrease in sum of diameters of target lesions, taking as reference baseline sum diameters or absence of a sufficient increase for PD, taking as reference the sum of lowest diameters during study.
Time Frame: At the end of study visit follow-up (during follow up period maximum of 39.8 months for Cases)
Population: Analysis population included all eligible participants whose data were observed in the study and who had attended at least end of study visit follow up. Here, "Overall number of participants analyzed" signifies participants evaluable for this outcome measure with non-missing values. This outcome measure was planned to be analyzed only in those participants with mRCC in CR.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 26
Participants
  Complete response | 7
  Partial response | 1
  Stabilized | 7
  Not applicable | 11

52. Primary Outcome: Duration of Treatment With First Line Sunitinib Till Progression: mRCC Participants With CR
Description: as for outcome 41
Time Frame: Sunitinib initiation (before inclusion, participants recruited for 3 years) till progression (follow up period maximum of 39.8 months for Cases)
Population: Analysis population included all eligible participants whose data were observed in the study and who had attended at least end of study visit follow up. Here, "Overall number of participants analyzed" signifies participants evaluable for this outcome measure. This outcome measure was planned to be analyzed only in those participants with mRCC in CR.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 11
Months | 24.5 (29.7)

53. Primary Outcome: Number of Participants Who Were Early Terminated: mRCC Participants With CR
Description: Participants who terminated study early were reported in this outcome measure.
Time Frame: From inclusion in the study till termination (during follow up period maximum of 39.8 months for Cases)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 35
Participants
  Yes | 2
  No | 33

54. Primary Outcome: Number of Participants Who Achieved Response: mRCC Participants With CR
Time Frame: At initiation of sunitinib (during follow up period maximum of 39.8 months for Cases)
Population: Data for this outcome measure was not collected, as there were less number of participants who had response.
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 0

55. Primary Outcome: Number of Participants Categorized According to Number of Subsequent Treatment Lines From Progression/Post Complete Remission: mRCC Participants With CR
Time Frame: At initiation of sunitinib (during follow up period maximum of 39.8 months for Cases)
Population: Data for this outcome measure was not collected, as there were less number of participants with an event.
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 0

56. Primary Outcome: Number of Participants Who Died: mRCC Participants With CR
Description: In this outcome measure, participants who died during the study were reported.
Time Frame: At initiation of sunitinib (during follow up period maximum of 39.8 months for Cases)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 35
Participants | 5

57. Primary Outcome: Progression Free Survival: mRCC Participants With CR
Description: PFS was based on Kaplan-Meier estimates. PFS was defined as time in months from start of treatment-to-treatment discontinuation due to disease progression as assessed by the investigator. PD: =>20% increase in sum of longest dimensions of lesions taking as a reference smallest sum of longest dimensions since treatment start or appearance of =>1 new lesions. Disease progression was determined from oncologic assessment data (where data meet the criteria for PD), or from death case report forms (CRFs). This outcome measure was analyzed by using Kaplan-Meier method.
Time Frame: At the end of the study (inclusion period was of 3 years and follow up period maximum of 39.8 months for Cases)
Population: as for outcome 17
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib: Complete Remission (Cases)
Number analyzed (Participants) | 35
Months | 69.4 [32.3 to NA] — Upper limit of 95% CI was not estimable, as there were less than 50% of participants with PFS.

58. Primary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. A serious AE was any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent or significant disability/ incapacity; congenital anomaly/birth defect and other important medical events.
Time Frame: During follow up period maximum of 39.8 months for Cases and 37 months for Controls
Population: Analysis population included all eligible participants whose data were observed in the study and who had attended at least one follow-up visit. Here, "Overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases) | Sunitinib: Non-Complete Remission (Control)
Number analyzed (Participants) | 35 | 41
Participants
  AEs | 32 | 41
  SAEs | 18 | 35

59. Primary Outcome: Number of Participants With Adverse Events and Serious Adverse Events Possibly Related to Drug Exposure
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study treatment, possibly considered related to the study treatment. A serious AE was any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent or significant disability/ incapacity; congenital anomaly/birth defect and other important medical events.
Time Frame: During follow up period maximum of 39.8 months for Cases and 37 months for Controls
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Complete Remission (Cases) | Sunitinib: Non-Complete Remission (Control)
Number analyzed (Participants) | 35 | 41
Participants
  AEs related to drug exposure | 15 | 41
  SAEs related to drug exposure | 3 | 21

60. Primary Outcome: Number of AEs According to Action Taken for the Study Treatment in Response to Those AEs
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Time Frame: During follow up period maximum of 39.8 months for Cases and 37 months for Controls
Population: as for outcome 4
Measure: Number; unit: Adverse events
Arm/Group | Sunitinib: Complete Remission (Cases) | Sunitinib: Non-Complete Remission (Control)
Number analyzed (Participants) | 32 | 41
Adverse events
  Drug interrupted (temporarily or permanent or dose delayed) | 16 | 72
  Dose reduced | 14 | 118
  Dose not changed | 83 | 330
  Unknown | 1 | 6
  Not applicable | 4 | 9
  Missing data | 2 | 6

61. Other Pre Specified Outcome: Number of Participants Categorized According to Types of Blood Biomarkers
Time Frame: During follow up period maximum of 39.8 months for Cases and 37 months for Controls
Population: Data was not available as the participating centers did not return the biological samples accordingly, to realize the analysis.
Arm/Group | Sunitinib: Complete Remission (Cases) | Sunitinib: Non-Complete Remission (Control)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: During follow up period maximum of 39.8 months for Cases and 37 months for Controls
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Sunitinib: Complete Remission (Cases) | Sunitinib: Non-Complete Remission (Control)
All-Cause Mortality (participants affected / at risk) | 5/35 | 20/41
Serious Adverse Events (participants affected / at risk) | 18/35 | 35/41
Other Adverse Events (participants affected / at risk) | 32/35 | 40/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib: Complete Remission (Cases) (N=35) | Sunitinib: Non-Complete Remission (Control) (N=41)
General physical health deterioration (General disorders) | 2 | 9
Disease evolution (General disorders) | 1 | 2
Asthenia (General disorders) | 0 | 2
Malaise (General disorders) | 0 | 2
Chest pain (General disorders) | 0 | 1
Death (General disorders) | 0 | 1
Drug ineffective (General disorders) | 0 | 1
Granuloma (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Oedema (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Mallory-weiss syndrome (Gastrointestinal disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1
Corona virus infection (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Pneumonia influenzal (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Superinfection bacterial (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Motor dysfunction (Nervous system disorders) | 1 | 1
Ataxia (Nervous system disorders) | 0 | 1
Balance disorder (Nervous system disorders) | 1 | 0
Dyskinesia (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Hemiplegia (Nervous system disorders) | 1 | 0
Neurological symptom (Nervous system disorders) | 0 | 1
Pachymeningitis (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Polycythaemia (Blood and lymphatic system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Ureteric stenosis (Renal and urinary disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Blood albumin decreased (Investigations) | 0 | 1
Blood catecholamines abnormal (Investigations) | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 2
Mental disorder (Psychiatric disorders) | 1 | 0
Breast disorder (Reproductive system and breast disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 1
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Medication error (Injury, poisoning and procedural complications) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Patient-device incompatibility (Product Issues) | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
Loss of personal independence in daily activities (Social circumstances) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib: Complete Remission (Cases) (N=35) | Sunitinib: Non-Complete Remission (Control) (N=41)
Asthenia (General disorders) | 10 | 25
Fatigue (General disorders) | 8 | 20
Mucosal inflammation (General disorders) | 3 | 25
Oedema peripheral (General disorders) | 3 | 9
Pyrexia (General disorders) | 1 | 11
General physical health deterioration (General disorders) | 2 | 7
Chest pain (General disorders) | 1 | 4
Gait disturbance (General disorders) | 1 | 3
Malaise (General disorders) | 1 | 3
Oedema (General disorders) | 2 | 2
Pain (General disorders) | 2 | 2
Face oedema (General disorders) | 0 | 3
Xerosis (General disorders) | 0 | 3
Chest discomfort (General disorders) | 0 | 2
Hyperthermia (General disorders) | 0 | 2
Impaired healing (General disorders) | 1 | 1
Mucosal haemorrhage (General disorders) | 0 | 2
Chills (General disorders) | 0 | 1
Feeling hot (General disorders) | 0 | 1
Injection site necrosis (General disorders) | 1 | 0
Injection site pain (General disorders) | 1 | 0
Injection site swelling (General disorders) | 0 | 1
Localised oedema (General disorders) | 1 | 0
Mucosal toxicity (General disorders) | 0 | 1
Thirst (General disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 14 | 32
Nausea (Gastrointestinal disorders) | 4 | 24
Vomiting (Gastrointestinal disorders) | 5 | 14
Abdominal pain upper (Gastrointestinal disorders) | 5 | 9
Constipation (Gastrointestinal disorders) | 3 | 11
Abdominal pain (Gastrointestinal disorders) | 4 | 7
Dyspepsia (Gastrointestinal disorders) | 2 | 8
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 7
Abdominal distension (Gastrointestinal disorders) | 1 | 5
Aphthous ulcer (Gastrointestinal disorders) | 0 | 6
Dysphagia (Gastrointestinal disorders) | 0 | 5
Haemorrhoids (Gastrointestinal disorders) | 1 | 4
Anorectal discomfort (Gastrointestinal disorders) | 0 | 4
Dry mouth (Gastrointestinal disorders) | 1 | 3
Gastric disorder (Gastrointestinal disorders) | 1 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 4
Stomatitis (Gastrointestinal disorders) | 1 | 3
Gingival bleeding (Gastrointestinal disorders) | 1 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 1 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 2
Reflux gastritis (Gastrointestinal disorders) | 0 | 2
Toothache (Gastrointestinal disorders) | 1 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal rigidity (Gastrointestinal disorders) | 0 | 1
Aerophagia (Gastrointestinal disorders) | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 1
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 | 1
Gingival recession (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Lip oedema (Gastrointestinal disorders) | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Rectal discharge (Gastrointestinal disorders) | 0 | 1
Tongue disorder (Gastrointestinal disorders) | 0 | 1
Tooth disorder (Gastrointestinal disorders) | 1 | 0
Varicose veins of abdominal wall (Gastrointestinal disorders) | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 | 23
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 11
Rash (Skin and subcutaneous tissue disorders) | 0 | 11
Erythema (Skin and subcutaneous tissue disorders) | 0 | 9
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 6
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 4
Skin toxicity (Skin and subcutaneous tissue disorders) | 3 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 2
Skin reaction (Skin and subcutaneous tissue disorders) | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0
Erythrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 | 1
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 | 1
Madarosis (Skin and subcutaneous tissue disorders) | 0 | 1
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Scar pain (Skin and subcutaneous tissue disorders) | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 1
Yellow skin (Skin and subcutaneous tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 4
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1
Clubbing (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint lock (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Torticollis (Musculoskeletal and connective tissue disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 4 | 14
Sciatica (Nervous system disorders) | 3 | 5
Headache (Nervous system disorders) | 1 | 6
Nervous system disorder (Nervous system disorders) | 2 | 2
Neuropathy peripheral (Nervous system disorders) | 2 | 2
Somnolence (Nervous system disorders) | 0 | 4
Ageusia (Nervous system disorders) | 0 | 3
Balance disorder (Nervous system disorders) | 0 | 2
Neuralgia (Nervous system disorders) | 1 | 1
Presyncope (Nervous system disorders) | 0 | 2
Apraxia (Nervous system disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 1
Burning sensation mucosal (Nervous system disorders) | 0 | 1
Cerebellar syndrome (Nervous system disorders) | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Hypogeusia (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Paraparesis (Nervous system disorders) | 1 | 0
Partial seizures with secondary generalisation (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Hypertension (Vascular disorders) | 12 | 19
Hypotension (Vascular disorders) | 3 | 3
Haematoma (Vascular disorders) | 0 | 3
Hot flush (Vascular disorders) | 2 | 1
Thrombosis (Vascular disorders) | 0 | 2
Aortic stenosis (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Varicose vein (Vascular disorders) | 0 | 1
Vena cava thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 8
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 8
Fungal infection (Infections and infestations) | 0 | 7
Bronchitis (Infections and infestations) | 2 | 4
Paronychia (Infections and infestations) | 0 | 3
Rhinitis (Infections and infestations) | 1 | 2
Conjunctivitis (Infections and infestations) | 0 | 2
Lung infection (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 2
Angular cheilitis (Infections and infestations) | 0 | 1
Bronchiolitis (Infections and infestations) | 1 | 0
Candida infection (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Genital herpes (Infections and infestations) | 0 | 1
Gingivitis (Infections and infestations) | 0 | 1
Hepatitis e (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Onychomycosis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Retinitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Spinal cord infection (Infections and infestations) | 0 | 1
Sputum purulent (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1
Vulvitis (Infections and infestations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 4 | 21
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2
Iron deficiency (Metabolism and nutrition disorders) | 1 | 2
Vitamin d deficiency (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Cell death (Metabolism and nutrition disorders) | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Food intolerance (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Vitamin b complex deficiency (Metabolism and nutrition disorders) | 1 | 0
Vitamin k deficiency (Metabolism and nutrition disorders) | 0 | 1
Weight fluctuation (Metabolism and nutrition disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 4 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 7
Neutropenia (Blood and lymphatic system disorders) | 3 | 2
Anaemia folate deficiency (Blood and lymphatic system disorders) | 0 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Macrocytosis (Blood and lymphatic system disorders) | 0 | 1
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 | 1
Weight decreased (Investigations) | 1 | 9
Blood thyroid stimulating hormone increased (Investigations) | 2 | 4
Breath sounds abnormal (Investigations) | 0 | 6
Blood creatinine increased (Investigations) | 0 | 3
Blood pressure abnormal (Investigations) | 1 | 2
Blood electrolytes abnormal (Investigations) | 0 | 1
Gastrointestinal stoma output increased (Investigations) | 0 | 1
Intestinal transit time decreased (Investigations) | 0 | 1
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 | 1
Oxygen saturation decreased (Investigations) | 1 | 0
Prostatic specific antigen increased (Investigations) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 5
Depressed mood (Psychiatric disorders) | 2 | 4
Depression (Psychiatric disorders) | 3 | 2
Confusional state (Psychiatric disorders) | 2 | 2
Sleep disorder (Psychiatric disorders) | 1 | 2
Mental disorder (Psychiatric disorders) | 0 | 2
Affective disorder (Psychiatric disorders) | 1 | 0
Anger (Psychiatric disorders) | 1 | 0
Body dysmorphic disorder (Psychiatric disorders) | 0 | 1
Depressive symptom (Psychiatric disorders) | 0 | 1
Hallucination, visual (Psychiatric disorders) | 0 | 1
Irritability (Psychiatric disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 6 | 9
Hyperthyroidism (Endocrine disorders) | 1 | 3
Thyroid mass (Endocrine disorders) | 1 | 1
Cushing's syndrome (Endocrine disorders) | 1 | 0
Thyroid disorder (Endocrine disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 4
Urinary tract disorder (Renal and urinary disorders) | 1 | 3
Dysuria (Renal and urinary disorders) | 1 | 2
Renal failure (Renal and urinary disorders) | 0 | 3
Acute kidney injury (Renal and urinary disorders) | 0 | 2
Proteinuria (Renal and urinary disorders) | 0 | 2
Renal impairment (Renal and urinary disorders) | 1 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 3
Breast pain (Reproductive system and breast disorders) | 0 | 2
Orchitis noninfective (Reproductive system and breast disorders) | 0 | 2
Scrotal inflammation (Reproductive system and breast disorders) | 0 | 2
Breast disorder (Reproductive system and breast disorders) | 1 | 0
Breast oedema (Reproductive system and breast disorders) | 0 | 1
Genital discomfort (Reproductive system and breast disorders) | 1 | 0
Genital disorder female (Reproductive system and breast disorders) | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Oligomenorrhoea (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Scrotal erythema (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal inflammation (Reproductive system and breast disorders) | 0 | 1
Eyelid oedema (Eye disorders) | 1 | 6
Diplopia (Eye disorders) | 0 | 3
Cataract (Eye disorders) | 1 | 1
Eye swelling (Eye disorders) | 0 | 2
Lacrimation increased (Eye disorders) | 0 | 2
Dry eye (Eye disorders) | 0 | 1
Eye disorder (Eye disorders) | 0 | 1
Eye pain (Eye disorders) | 0 | 1
Ocular discomfort (Eye disorders) | 1 | 0
Periorbital oedema (Eye disorders) | 1 | 0
Uveitis (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Injury (Injury, poisoning and procedural complications) | 2 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 2 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Radiation necrosis (Injury, poisoning and procedural complications) | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 1
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Jaundice (Hepatobiliary disorders) | 2 | 7
Hepatocellular injury (Hepatobiliary disorders) | 0 | 3
Hepatic pain (Hepatobiliary disorders) | 0 | 1
Ocular icterus (Hepatobiliary disorders) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Retroperitoneal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Extrasystoles (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 3
Hyperacusis (Ear and labyrinth disorders) | 0 | 1
Amyloidosis (Immune system disorders) | 1 | 0
Sarcoidosis (Immune system disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 1
Patient-device incompatibility (Product Issues) | 0 | 1
Appendicectomy (Surgical and medical procedures) | 0 | 1
Psychiatric decompensation (Psychiatric disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/52/NCT01934452/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-30): https://cdn.clinicaltrials.gov/large-docs/52/NCT01934452/SAP_001.pdf